CLINICAL TRIAL: NCT03291002
Title: Phase I Study of Intratumoral CV8102 in Patients With Advanced Melanoma, Squamous Cell Carcinoma of the Skin, Squamous Cell Carcinoma of the Head and Neck, or Adenoid Cystic Carcinoma
Brief Title: Study of Intratumoral CV8102 in cMEL, cSCC, hnSCC, and ACC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CureVac (Industry)
Collaborators: Syneos Health (Other); Cromos Pharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-8102-008
Record Dates: First submitted 2017-09-15; First posted 2017-09-25 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Melanoma (Skin); Squamous Cell Carcinoma of the Skin; Carcinoma, Squamous Cell of Head and Neck; Carcinoma, Adenoid Cystic
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Intervention Model Description: Open-label, cohort-based, dose escalation and expansion study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Dose escalation of CV8102
  Interventions: Biological: CV8102
- Cohort B (Experimental): Optional expansion cohorts of CV8102
  Interventions: Biological: CV8102
- Cohort C (Experimental): Dose escalation of CV8102 + anti-PD-1 therapy
  Interventions: Biological: CV8102 + anti-PD-1 therapy
- Cohort D (Experimental): Optional expansion of CV8102 + anti-PD-1 therapy
  Interventions: Biological: CV8102 + anti-PD-1 therapy

INTERVENTIONS:
Biological: CV8102 — CV8102 alone
  Arms: Cohort A; Cohort B
Biological: CV8102 + anti-PD-1 therapy — CV8102 in combination with standard of care anti-PD-1 therapy
  Arms: Cohort C; Cohort D

SUMMARY:
This study evaluates intratumoral administration of CV8102 in patients with advanced melanoma, squamous cell carcinoma of the skin, squamous cell carcinoma of the head and neck, or adenoid cystic carcinoma.

Patients will receive CV8102 as single agent or in combination with SoC anti-PD-1 therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients enrolled into Cohorts A and B (single agent CV8102) must have:

   * histologically confirmed advanced cutaneous melanoma, cutaneous squamous cell carcinoma, head and neck squamous cell carcinoma, or adenoid cystic carcinoma with documented disease progression
   * not amenable to surgical resection or locoregional radiation therapy with curative intent
   * at least 1 line of anti-cancer therapy for advanced disease (except adenoid cystic carcinoma) and documented Progression
   * cutaneous melanoma Cohort B3: Willing to undergo baseline and post-baseline biopsy of the lesion which is to be injected
2. Patients enrolled into Cohort C (CV8102 in combination with anti-PD-1 therapy) must have

   * histologically confirmed advanced cMEL or hnSCC
   * indication for anti-PD-1 therapy or currently receiving anti-PD-1 therapy with stable of slowly progressing disease after at last 8 weeks (hnSCC) or 12 weeks (cMEL) of anti-PD-1 therapy prior to Day 1
3. Patients enrolled into Cohort D1 (CV8102 in combination with anti-PD-1 therapy) must have

   * histologically confirmed advanced cMEL
   * either anti-PD-1 naive patients with indication for anti-PD-1 therapy (Cohort D1a) or patients refractory to anti-PD-1 therapy (Cohort D1b)
   * Presence of measurable lesion(s) according to RECIST 1.1, not intended for injection
   * Willing to undergo tumor biopsies at specific timepoints (Cohort D1a: baseline; Cohort D1b baseline and post-baseline biopsy of the injected lesion - only for selected sites)
4. Patients enrolled into Cohort D2 (CV8102 in combination with anti-PD-1 therapy) must have

   * histologically confirmed advanced hnSCC
   * indication for treatment with first-line pembrolizumab (patients naive to anti-PD-1/anti-PD-L1)
   * PD-L1 combined positive score ≥ 1% according to local practice
5. Presence of at least one injectable tumor lesion that is measurable according to RECIST 1.1
6. Recovered from prior toxicities to CTCAE grade ≤ 1 or grade ≤ 2
7. Resolution of CPI-related adverse effects, if applicable (including irAEs) back to CTCAE grade 0/1
8. ECOG PS 0 or 1
9. 18 years of age or older
10. Adequate hematologic, renal, hepatic and coagulation function
11. Use of effective contraception

Key Exclusion Criteria:

1. Rapidly progressing multi-focal metastatic or acutely life threatening disease
2. Prior use of topical/localTLR-7/8 agonists within the past 6 months
3. Clinically active central nervous system metastases and/or carcinomatous meningitis (patients with stable brain metastases are eligible)
4. Ocular and mucosal melanoma
5. Prior anti-cancer therapy within specified time-periods depending on the indication
6. Tumor lesions that are to be injected close to major blood vessels or nerves, or whose injection could potentially result in clinical adverse effects if post-treatment tumor swelling or inflammation were to occur
7. Lesions that are to be injected in previously irradiated areas unless progressive tumor growth has been demonstrated (no prior irradiation of injected lesions on patients with melanoma)
8. History of active coagulation or bleeding disorder or need for ongoing therapeutic anticoagulation that cannot be safely interrupted at th etime of IT injection or biopsy du eto Underlying medical conditions; patients with melanoma and cutaneous squamous cell carcinoma with controlled oral anticoagulation are eligible
9. Treatment with any investigational anticancer agent within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug or planned during the study
10. Acute hypophysitis or endocrinopathies that are not adequately controlled by hormonal replacement therapy or thyreostatic treatment
11. Use of immune modulating drugs or immunologically active topical therapies within 28 days of administration of the first dose of study drug
12. Chronic systemic immunosuppressive therapy including chronic corticosteroids within 28 days of the first dose of study drug (except physiological maintenance/replacement steroid doses, topical steroids outside the injected lesion or inhaled steroids); patients are eligible if steroid requirement is < 10 mg/day of prednisone (or equivalent) for at least 2 weeks
13. History of active autoimmune disease requiring immunosuppressive medication (except Vitiligo and except CPI-mediated irAEs)
14. Known hematologic malignancy or malignant primary solid tumor that have occured or reoccurred within the previous 5 years
15. Recent thromboembolic complications, or clinically significant cardiovascular disease, or any other uncontrolled illness that would pose a risk to patient safety
16. Severe infection or acute inflammatory state
17. Seropositivity for human immunodeficiency virus (HIV), hepatitis B virus (HBV) surface antigen (except in previously vaccinated patients) or hepatitis C virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Dose determination for dose escalation cohorts | 2 weeks
  * Maximum tolerated dose (MTD) and recommended dose (RD), respectively, for CV8102 alone
  * MTD and recommended combination dose (RCD) for CV8102 in combination with the standard dose of an anti-PD-1 antagonist
Incidence of treatment related (Serious) Adverse Events (Tolerability and Safety profile) | up to 12 months (end of study)
  • Tolerability and safety profile of CV8102 alone and in combination with anti-PD-1 antagonists

SECONDARY OUTCOMES:
Tumor response | up to 12 months (end of study)
  • Anti-tumor activity of CV8102 per irRECIST and RECIST 1.1
Disease status | 6 months
  • Tumor Assessment
Tumor response | up to 12 months (end of study)
  • Extent of tumor response at injected and non-injected lesions, if applicable
Survival | up to 12 months (end of study)
  • Survival time

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eigentler, Prof. Dr., Principal Investigator — thomas.eigentler@charite.de
Locations (22):
- Austria (2):
  - Medical University of Graz, Graz
  - Universitätsklinik für Dermatologie der Paracelsus medizinischen Privatuniversität Salzburg, Salzburg
- France (2):
  - Hôpital Saint Louis, Paris
  - Institut Gustave Roussy, Paris
- Germany (9):
  - Charité Benjamin Franklin, Berlin
  - Medizinische Klinik III, Universitätsklinikum Bonn, Hämatologie, Immunonkologie und Rheumatologie, Bonn
  - Elbe-Klinikum-Buxtehude, Hautkrebszentrum, Buxtehude
  - Universitätsklinikum Erlangen,Hautklinik, Internistisches Zentrum (INZ), Erlangen
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Klinik für Dermatologie, Allergologie und Venerologie, Lübeck
  - Fachklinik Hornheide, Münster
  - Universitätsklinikum Münster, Klinik für Hautkrankheiten, ZiD- Zentrum für innovative Dermatologie, Münster
  - Universitäts-Hautklinik, Abtl. Dermatologische Onkologie, Tübingen
- Russia (4):
  - Center for Personalized Oncology, I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation, Moscow
  - FSBI "National Medical Research Center of Oncology n.a. N.N. Blokhin" of the Ministry of Healthcare of the Russian Federation, Moscow
  - FSBI "National Medical Research Oncology Center n.a. N.N. Petrov, Saint Petersburg
  - Saint-Petersburg State University, Clinic of advanced medical technologies n. a. Nicolay I. Pirogov., Saint Petersburg
- Spain (5):
  - Hospital Duran i Reynals - Institut Catala dOncologia ICO, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marqus de Valdecilla Santander, Santander

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eigentler T, Thomas I, Samoylenko I, Erdmann M, Heinzerling L, Ochsenreither S, Krauss J, Oberoi A, Robert C, Lebbe C, Martin-Liberal J, Koch L, Richtig E, Terheyden P, Weishaupt C, Mohr P, Semiletova Y, Perez CL, Brossart P, Bauernfeind FG, Fluck M, Poltoratskiy A, Sekacheva M, Soria A, Schmitt-Bormann B, Gonzalez M, Hess J, Wengenmayer P, Seibel T, Koch SD, Quintini G, Codo P, Falk M, Schonborn-Kellenberger O, Gnad-Vogt U. Phase I study of intratumoral administration of CV8102 in patients with advanced melanoma, squamous cell carcinoma of the skin, squamous cell carcinoma of the head and neck, or adenoid cystic carcinoma. J Immunother Cancer. 2025 Feb 4;13(2):e009352. doi: 10.1136/jitc-2024-009352. PMID 39904560
- [Derived] Lutz J, Meister M, Habbeddine M, Fiedler K, Kowalczyk A, Heidenreich R. Local immunotherapy with the RNA-based immune stimulator CV8102 induces substantial anti-tumor responses and enhances checkpoint inhibitor activity. Cancer Immunol Immunother. 2023 May;72(5):1075-1087. doi: 10.1007/s00262-022-03311-4. Epub 2022 Nov 2. PMID 36319717